CLINICAL TRIAL: NCT00731068
Title: PRP as a Treatment for ACHILLES Tendon Tears - Randomized-Double-Blind-Placebo Control Trail
Brief Title: Platelet Rich Plasma (PRP) as a Treatment for ACHILLES Tendon Tears
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2000; MeirMc07om0090CTIL
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Achilles Tendon Tear
Keywords: Achilles tendon
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): PRGF
  Interventions: Biological: PRGF
- 2 (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: PRGF — injection of 6cc into injured area of tendon
  Other Names: platelet-derived preparation rich in growth factors
  Arms: 1
Biological: placebo — injection of 6 cc of saline into injured area
  Other Names: saline 0.9% nacl
  Arms: 2

SUMMARY:
To review the influence of patient derived PRGF on the healing process of Achilles tendon after a surgical correction of a complete tear.

DETAILED DESCRIPTION:
Autologous platelet-rich matrices may aid in post surgical patients by promoting and accelerating tissue healing because of the release of growth factors including transforming growth factor (TGF)-beta1 and platelet-derived growth factor (PDGF) from platelet alpha-granules.

ELIGIBILITY:
Inclusion Criteria:

* A complete tear of Achilles tendon
* Age 18-50 years old

Exclusion Criteria:

* under 18 year of age
* pregnancy
* physical or mental disabilities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
improvement of symptoms / disease progress | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mei Dan, Dr, Principal Investigator — Meir Medical Center